CLINICAL TRIAL: NCT02624778
Title: A Single- and Multiple-Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Intravenous Doses of LY3002813 in Patients With Mild Cognitive Impairment Due to Alzheimer's Disease or Mild to Moderate Alzheimer's Disease
Brief Title: A Study of LY3002813 in Participants With Memory Damage Due to Alzheimer's Disease (AD) or AD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 16233; I5T-MC-AACD (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-12-04; First posted 2015-12-08 (Estimated); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Part A: Placebo Single Dose (SD) (Placebo Comparator): Participants received single intravenous (IV) dose of placebo.
  Interventions: Drug: Placebo
- Part A: 10 Milligram Per Kilogram (mg/kg) LY3002813 SD (Experimental): Participants received single IV dose of 10 mg/kg LY3002813.
  Interventions: Biological: LY3002813
- Part A: 20 mg/kg LY3002813 SD (Experimental): Participants received single IV dose of 20 mg/kg LY3002813.
  Interventions: Biological: LY3002813
- Part A: 40 mg/kg LY3002813 SD (Experimental): Participants received single IV dose of 40 mg/kg LY3002813.
  Interventions: Biological: LY3002813
- Part B: Placebo Q2W (Placebo Comparator): Participants received multiple IV dose of placebo every 2 weeks (Q2W) for 24 weeks.
  Interventions: Drug: Placebo
- Part B: 10 mg/kg LY3002813 Q2W (Experimental): Participants received multiple IV dose of 10 mg/kg LY3002813 Q2W for 24 weeks.
  Interventions: Biological: LY3002813
- Part C: Placebo Q4W (Placebo Comparator): Participants received multiple IV dose of placebo every 4 weeks (Q4W) for 72 weeks.
  Interventions: Drug: Placebo
- Part C:10 mg/kg LY3002813 Q4W (Experimental): Participants received multiple IV dose of 10 mg/kg LY3002813 Q4W for 72 weeks.
  Interventions: Biological: LY3002813
- Part C:20 mg/kg LY3002813 Q4W (Experimental): Participants received multiple IV dose of 20 mg/kg LY3002813 Q4W for 72 weeks.
  Interventions: Biological: LY3002813

INTERVENTIONS:
Biological: LY3002813 — Administered IV
  Arms: Part A: 10 Milligram Per Kilogram (mg/kg) LY3002813 SD; Part A: 20 mg/kg LY3002813 SD; Part A: 40 mg/kg LY3002813 SD; Part B: 10 mg/kg LY3002813 Q2W; Part C:10 mg/kg LY3002813 Q4W; Part C:20 mg/kg LY3002813 Q4W
Drug: Placebo — Administered IV
  Arms: Part A: Placebo Single Dose (SD); Part B: Placebo Q2W; Part C: Placebo Q4W

SUMMARY:
The study will evaluate the effect of LY3002813 on brain scans. The study will evaluate the safety of LY3002813 by looking at adverse events (side effects). The study will also look at the effect the body has on LY3002813. Study participants will have mild cognitive impairment (MCI) due to AD or mild to moderate AD.

The study involves 3 parts.

* Part A in which participants will receive a single dose of LY3002813 or placebo (no drug).
* Part B in which participants will receive multiple doses of LY3002813 or placebo for 24 weeks.
* Part C in which participants will receive multiple doses of LY3002813 or placebo for up to 72 weeks.

Drug will be given as an intravenous infusion (injection into a vein). For Parts A, B and C, the study will last approximately 72 weeks, not including screening of approximately 56 days. The study is for research purposes only and is not intended to treat any medical condition.

ELIGIBILITY:
Inclusion Criteria:

* Present with mild cognitive impairment (MCI) due to Alzheimer's disease (AD) or mild-to-moderate AD
* Men or nonfertile women, at least 50 years of age. Nonfertile is defined as hysterectomy and/or bilateral oophorectomy, or amenorrhea for at least 1 year
* Have up to 2 partners who will provide a separate written informed consent to participate
* Have adequate vision and hearing for neuropsychological testing in the opinion of the investigator
* Positive florbetapir scan

Exclusion Criteria:

* Do not have up to 2 reliable partners who are in frequent contact with the participant, who will accompany the participant to the office and/or be available by telephone at designated times, and will monitor administration of prescribed medications
* Are being monitored for radiation due to occupational exposure to ionized radiation, or exposure to ionizing radiation within last 12 months from an investigational study
* History of intracranial hemorrhage, cerebrovascular aneurysm or arteriovenous malformation, or carotid artery occlusion, or stroke or epilepsy
* Have any contraindications for magnetic resonance imaging (MRI) studies, including claustrophobia, the presence of contraindicated metal (ferromagnetic) implants, cardiac pacemaker
* Have allergies to humanized monoclonal antibodies, including proteins and diphenhydramine, epinephrine, and methylprednisolone
* Have gamma globulin therapy within the last year
* Previously dosed in any other study investigating active immunization against amyloid beta (Aβ)
* Previously dosed in any other study investigating passive immunization against Aβ within the last 6 months
* Have current serious or unstable illnesses

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- United States (6):
  - Brain Matters Research, Delray Beach, Florida
  - Compass Research, Orlando, Florida
  - Compass Research, The Villages, Florida
  - SNBL Clinical Pharmacology Center Inc, Baltimore, Maryland
  - St. Louis Clinical Trials, LC, St Louis, Missouri
  - PRA Health Sciences, Salt Lake City, Utah
- Japan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shinjuku-Ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Shinjuku-Ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Sumida-ku

REFERENCES:
- See also: Click here for more information about this study: A Study of LY3002813 in Participants With Memory Damage Due to Alzheimer's Disease (AD) — http://www.lillytrialguide.com/EN-us/studies/alzheimer's/aacd

RESULTS

PARTICIPANT FLOW:
Groups:
- Part B: Placebo Q2W: Participants received multiple IV doses of placebo every 2 weeks (Q2W) for 24 weeks.
- Part B: 10 mg/kg LY3002813 Q2W: Participants received multiple IV doses of 10 mg/kg LY3002813 Q2W for 24 weeks.
- Part C: Placebo Q4W: Participants received multiple IV doses of placebo every 4 weeks (Q4W) for 72 weeks.
- Part C:10 mg/kg LY3002813 Q4W: Participants received multiple IV doses of 10 mg/kg LY3002813 Q4W for 72 weeks.
- Part C:20 mg/kg LY3002813 Q4W: Participants received multiple IV doses of 20 mg/kg LY3002813 Q4W for 72 weeks.
Period: Overall Study
Arm/Group | Part A: Placebo Single Dose (SD) | Part A: 10 Milligram Per Kilogram (mg/kg) LY3002813 SD | Part A: 20 mg/kg LY3002813 SD | Part A: 40 mg/kg LY3002813 SD | Part B: Placebo Q2W | Part B: 10 mg/kg LY3002813 Q2W | Part C: Placebo Q4W | Part C:10 mg/kg LY3002813 Q4W | Part C:20 mg/kg LY3002813 Q4W
Started | 7 | 7 | 7 | 4 | 3 | 10 | 5 | 8 | 10
Received at Least 1 Dose of Study Drug | 7 | 7 | 7 | 4 | 3 | 10 | 5 | 8 | 10
Completed | 7 | 6 | 6 | 4 | 3 | 9 | 3 | 4 | 4
Not Completed | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 4 | 6
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Part A: 10 mg/kg LY3002813 SD: Participants received single IV dose of 10 mg/kg LY3002813.
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo Single Dose (SD) | Part A: 10 mg/kg LY3002813 SD | Part A: 20 mg/kg LY3002813 SD | Part A: 40 mg/kg LY3002813 SD | Part B: Placebo Q2W | Part B: 10 mg/kg LY3002813 Q2W | Part C: Placebo Q4W | Part C:10 mg/kg LY3002813 Q4W | Part C:20 mg/kg LY3002813 Q4W | Total
Number analyzed (Participants) | 7 | 7 | 7 | 4 | 3 | 10 | 5 | 8 | 10 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.6 (7.7) | 78.3 (8.4) | 75.6 (6.4) | 75.3 (6.7) | 65.7 (4.9) | 66.8 (8.6) | 72.6 (12.2) | 73.0 (7.8) | 71.7 (9.2) | 73.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 3 | 2 | 2 | 4 | 3 | 4 | 6 | 34
  Male | 1 | 3 | 4 | 2 | 1 | 6 | 2 | 4 | 4 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 7 | 7 | 7 | 4 | 3 | 9 | 5 | 8 | 9 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 1 | 2 | 1 | 3 | 2 | 3 | 2 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
  White | 4 | 5 | 6 | 1 | 2 | 7 | 3 | 5 | 7 | 40
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 6 | 2 | 2 | 7 | 3 | 5 | 8 | 43
  Japan | 2 | 2 | 1 | 2 | 1 | 3 | 2 | 3 | 2 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Florbetapir Positron Emission Tomography (PET) Scan Standard Uptake Value Ratio (SUVr)
Description: Florbetapir PET imaging was used to confirm the presence of amyloid pathology consistent with AD. Change from baseline was done to test the hypothesis that amyloid burden was reduced in participants in the treatment group. The change from baseline to the postbaseline visit of the composite summary standard uptake value ratio of florbetapir F18 was calculated. Least square (LS) mean value was controlled for baseline value, baseline age, pooled investigator, treatment and visit. The composite summary measure is an unweighted average of the 6 smaller regions (anterior cingulate, frontal medial orbital, parietal, posterior cingulate, precuneus, and temporal) normalized to whole cerebellum or subject-specific white matter.
Time Frame: Baseline, Week 72
Population: All randomized participants who received at least 1 dose of study drug and had baseline and post baseline scan data.
Measure: Least Squares Mean (Standard Error); unit: standard uptake value ratio (SUVr)
Groups:
- Part A,B and C: Placebo: Participants received single or multiple IV doses of placebo.
Arm/Group | Part A,B and C: Placebo | Part A: 10 mg/kg LY3002813 SD | Part A: 20 mg/kg LY3002813 SD | Part A: 40 mg/kg LY3002813 SD | Part B: 10 mg/kg LY3002813 Q2W | Part C:10 mg/kg LY3002813 Q4W | Part C:20 mg/kg LY3002813 Q4W
Number analyzed (Participants) | 11 | 6 | 6 | 1 | 9 | 4 | 4
standard uptake value ratio (SUVr) | -0.050 (0.04) | -0.122 (0.06) | -0.183 (0.06) | -0.255 (0.10) | -0.305 (0.05) | -0.419 (0.06) | -0.379 (0.05)
Statistical Analysis 1: Comparison: Part A,B and C: Placebo vs Part A: 10 mg/kg LY3002813 SD; Test type: Superiority; p = 0.309, Mixed Models Analysis; LS Mean = -0.071, 95% CI 2-sided [-0.21 to 0.07], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Part A,B and C: Placebo vs Part A: 20 mg/kg LY3002813 SD; Test type: Superiority; p = 0.061, Mixed Models Analysis; LS Mean = -0.133, 95% CI 2-sided [-0.27 to 0.01], Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Part A,B and C: Placebo vs Part A: 40 mg/kg LY3002813 SD; Test type: Superiority; p = 0.053, Mixed Models Analysis; LS Mean = -0.205, 95% CI 2-sided [-0.41 to 0.00], Standard Error of Mean 0.10
Statistical Analysis 4: Comparison: Part A,B and C: Placebo vs Part B: 10 mg/kg LY3002813 Q2W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean = -0.255, 95% CI 2-sided [-0.38 to -0.13], Standard Error of Mean 0.06
Statistical Analysis 5: Comparison: Part A,B and C: Placebo vs Part C:10 mg/kg LY3002813 Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean = -0.369, 95% CI 2-sided [-0.51 to -0.23], Standard Error of Mean 0.07
Statistical Analysis 6: Comparison: Part A,B and C: Placebo vs Part C:20 mg/kg LY3002813 Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean = -0.329, 95% CI 2-sided [-0.46 to -0.20], Standard Error of Mean 0.07

2. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-tlast)] in Part A
Description: Area under the curve from time zero to last quantifiable concentration [AUC (0-tlast)] at day 1 was reported.
Time Frame: Predose, end of infusion, 3, 24 and 48 hours postdose
Population: All randomized participants from part A who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter(μg*hr/mL)
Arm/Group | Part A: 10 mg/kg LY3002813 SD | Part A: 20 mg/kg LY3002813 SD | Part A: 40 mg/kg LY3002813 SD
Number analyzed (Participants) | 7 | 7 | 4
microgram*hour per milliliter(μg*hr/mL) | 25700 (20) | 59400 (19) | 110000 (32)

3. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Curve Versus Time at a Dosing Interval (AUCtau) at Day 1 of LY3002813 in Part B and Part C
Description: Area under the concentration versus time curve during one dosing interval at day 1 was reported.
Time Frame: Predose, end of infusion, 3, 24, 48 and 72 hours postdose
Population: All randomized participants from part B and part C who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (μg*hr/mL)
Arm/Group | Part B: 10 mg/kg LY3002813 Q2W | Part C:10 mg/kg LY3002813 Q4W | Part C:20 mg/kg LY3002813 Q4W
Number analyzed (Participants) | 9 | 8 | 10
microgram*hour per milliliter (μg*hr/mL) | 23000 (22) | 32900 (35) | 58900 (22)

4. Secondary Outcome: PK:Area Under the Concentration Curve Versus Time at a Dosing Interval at Steady State (AUCtau,ss) of LY3002813 in Part B and C
Description: AUCtau of LY3002813 at steady state (Day 127 [10 mg/kg Q2W] for part B and Day 141 [10 mg/kg and 20 mg/kg Q4W]) for Part C following multiple dose administration of LY3002813 was evaluated.
Time Frame: Part B (Day 127): predose, end of infusion, 3, 24, 48 and 72 hours postdose; Part C (Day 141): predose, end of infusion, 3, 24, 48 and 72 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*hr/mL
Arm/Group | Part B: 10 mg/kg LY3002813 Q2W | Part C:10 mg/kg LY3002813 Q4W | Part C:20 mg/kg LY3002813 Q4W
Number analyzed (Participants) | 4 | 6 | 7
μg*hr/mL | 29700 (68) | 35800 (61) | 68400 (37)

5. Secondary Outcome: PK: Maximum Serum Concentration (Cmax) of LY3002813 at Day 1 of LY3002813
Description: Maximum serum concentration of LY3002813 during one dosing interval at day 1 was reported.
Time Frame: Part A: Predose, end of infusion, 3, 24 and 48 hours postdose; Part B and C: Predose, end of infusion, 3, 24, 48 and 72 hours postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (μg/mL)
Arm/Group | Part A: 10 mg/kg LY3002813 SD | Part A: 20 mg/kg LY3002813 SD | Part A: 40 mg/kg LY3002813 SD | Part B: 10 mg/kg LY3002813 Q2W | Part C:10 mg/kg LY3002813 Q4W | Part C:20 mg/kg LY3002813 Q4W
Number analyzed (Participants) | 7 | 7 | 4 | 9 | 8 | 10
microgram per milliliter (μg/mL) | 196 (17) | 413 (17) | 910 (15) | 223 (19) | 252 (31) | 564 (26)

6. Secondary Outcome: PK: Maximum Serum Concentration (Cmax) of LY3002813 at Steady State of LY3002813 in Part B and C
Description: Cmax of LY3002813 at steady state (Day 127 [10 mg/kg Q2W] for part B and Day 141 [10 mg/kg and 20 mg/kg Q4W]) for Part C following multiple dose administration of LY3002813 was evaluated.
Time Frame: as for outcome 4
Population: All randomized participants from part B and C who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Part B: 10 mg/kg LY3002813 Q2W | Part C:10 mg/kg LY3002813 Q4W | Part C:20 mg/kg LY3002813 Q4W
Number analyzed (Participants) | 4 | 6 | 7
μg/mL | 273 (23) | 366 (44) | 598 (23)

7. Secondary Outcome: Percentage of Participants With Treatment-Emergent Anti-Drug Antibodies (TE-ADAs) to LY3002813
Description: Blood samples were tested to determine if a participant reacted to LY3002813 by producing anti-LY3002813 antibodies. Samples were identified as TE-ADAs if the post-treatment sample had an increase of at least 4 fold in titer from pre-treatment values. If the pre-treatment value was not detected or was not present, a 1:20 post-treatment titer was required to indicate treatment emergence. The percentage of participants with TE ADA was calculated as: (the number of participants with TE ADA / total number of participants with at least 1 post-treatment immunogenicity sample analyzed)*100.
Time Frame: Predose up to Day 589
Population: All randomized participants who received at least one dose of study drug & had least one non-missing test result for ADA for each of the baseline period and the post-baseline period.
Measure: Number; unit: percentage of participants
Groups:
- 10 mg/kg LY3002813 IV SD: Participants received single IV dose of 10 mg/kg LY3002813.
- 20 mg/kg LY3002813 IV SD: Participants received single IV dose of 20 mg/kg LY3002813.
- 40 mg/kg LY3002813 IV SD: Participants received single IV dose of 40 mg/kg LY3002813.
- 10 mg/kg LY3002813 IV Q2W: Participants received multiple IV doses of 10 mg/kg LY3002813 Q2W for 24 weeks.
- 10 mg/kg LY3002813 IV Q4W: Participants received multiple IV doses of 10 mg/kg LY3002813 Q4W for 72 weeks.
- 20 mg/kg LY3002813 IV Q4W: Participants received multiple IV doses of 20 mg/kg LY3002813 Q4W for 72 weeks.
Arm/Group | Part A,B and C: Placebo | 10 mg/kg LY3002813 IV SD | 20 mg/kg LY3002813 IV SD | 40 mg/kg LY3002813 IV SD | 10 mg/kg LY3002813 IV Q2W | 10 mg/kg LY3002813 IV Q4W | 20 mg/kg LY3002813 IV Q4W
Number analyzed (Participants) | 15 | 7 | 7 | 4 | 10 | 8 | 10
percentage of participants | 13.3 | 85.7 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

ADVERSE EVENTS:
Time Frame: Baseline Upto 584 Days
Description: All randomized participants who received at least 1 dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Part A: Placebo SD: Participants received single IV dose of placebo.
- Part B: Placebo Q2W: Participants received multiple IV doses of placebo Q2W for 24 weeks.
- Part C: Placebo Q4W: Participants received multiple IV doses of placebo Q4W for 72 weeks.
Arm/Group | Part A: Placebo SD | Part A: 10 mg/kg LY3002813 SD | Part A: 20 mg/kg LY3002813 SD | Part A: 40 mg/kg LY3002813 SD | Part B: Placebo Q2W | Part B: 10 mg/kg LY3002813 Q2W | Part C: Placebo Q4W | Part C:10 mg/kg LY3002813 Q4W | Part C:20 mg/kg LY3002813 Q4W
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7 | 0/4 | 0/3 | 0/10 | 1/5 | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/7 | 0/7 | 0/7 | 0/4 | 0/3 | 0/10 | 1/5 | 1/8 | 2/10
Other Adverse Events (participants affected / at risk) | 5/7 | 7/7 | 6/7 | 4/4 | 2/3 | 10/10 | 4/5 | 8/8 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A: Placebo SD (N=7) | Part A: 10 mg/kg LY3002813 SD (N=7) | Part A: 20 mg/kg LY3002813 SD (N=7) | Part A: 40 mg/kg LY3002813 SD (N=4) | Part B: Placebo Q2W (N=3) | Part B: 10 mg/kg LY3002813 Q2W (N=10) | Part C: Placebo Q4W (N=5) | Part C:10 mg/kg LY3002813 Q4W (N=8) | Part C:20 mg/kg LY3002813 Q4W (N=10)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased activity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/6 (1) | 0/4 (0) | 0/3 (0) | 0/2 (0) | 0/2 (0) | 0/4 (0) | 0/3 (0) | 0/4 (0) | 0/6 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anger (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A: Placebo SD (N=7) | Part A: 10 mg/kg LY3002813 SD (N=7) | Part A: 20 mg/kg LY3002813 SD (N=7) | Part A: 40 mg/kg LY3002813 SD (N=4) | Part B: Placebo Q2W (N=3) | Part B: 10 mg/kg LY3002813 Q2W (N=10) | Part C: Placebo Q4W (N=5) | Part C:10 mg/kg LY3002813 Q4W (N=8) | Part C:20 mg/kg LY3002813 Q4W (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodal rhythm (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased activity (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatophytosis of nail (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural anxiety (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (3)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased vibratory sense (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dementia alzheimer's type (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness exertional (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (4) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superficial siderosis of central nervous system (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 2 (2)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anger (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delusional perception (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressive symptom (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersomnia related to another mental condition (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Sterile pyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1/6 (1) | 0/4 (0) | 0/3 (0) | 0/2 (0) | 1/2 (1) | 0/4 (0) | 0/3 (0) | 0/4 (0) | 0/6 (0)
Breast pain (Reproductive system and breast disorders) | 0/6 (0) | 0/4 (0) | 0/3 (0) | 0/2 (0) | 0/2 (0) | 1/4 (1) | 0/3 (0) | 0/4 (0) | 0/6 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systolic hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor cannot use results communications, embargo communications regarding trial results for at least 5 years from the date of disclosure.

DOCUMENTS (2):
  • Study Protocol (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT02624778/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT02624778/SAP_001.pdf